CLINICAL TRIAL: NCT01401868
Title: Phase I Open Label Dose Escalation Study of the Safety and Pharmacokinetics of ME-143 as a Single Agent in Patients With Refractory Solid Tumors
Brief Title: Phase I Dose Escalation Study of the Safety and Pharmacokinetics of ME-143 Single Agent for Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MEI Pharma, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-143-001
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Solid Tumors
Keywords: solid tumor; recurrent; advanced; metastatic
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — ME-143; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): dose escalation
  Interventions: Drug: ME-143

INTERVENTIONS:
Drug: ME-143 — experimental drug, dose escalation with 4 dose cohorts of 2.5 mg/kg, 5 mg/kg, 10 mg/kg, 20 mg/kg; Cycle 1 is 3 weekly IV infusions on Days 1, 8 and 15. If either the 10 mg/kg or 20 mg/kg dose levels are not tolerable, a 7.5 mg/kg or a 15 mg/kg dose level will be evaluated. After safety assessment, if there is clinical benefit, weekly dosing may continue until withdrawal.
  Once the highest tolerated dose has been determined, patients will be enrolled to receive IV infusions 2-days per week. Cycle 1 at the highest dose level is 3 weekly IV infusions on Days 1, 2, 8, 9, 15 and 16. After safety assessment, if there is clinical benefit, weekly dosing may continue until withdrawal.
  Other Names: open label; single agent

SUMMARY:
The purpose of this study is to determine the tolerability of ME-143, find the maximum tolerated dose, and the safety profile in patients with refractory solid tumors.

DETAILED DESCRIPTION:
The purpose of this study is to determine the tolerability of ME-143, find the maximum tolerated dose, dose limiting toxicities, and the safety profile in patients with refractory solid tumors. In addition, the study is planned to characterize the pharmacokinetic profile of ME-143 and describe any clinical anti-tumor activity observed in patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Male or female ≥18 years of age
* Histologic or cytologic confirmed locally advanced or metastatic cancer that has no standard therapeutic alternatives.
* ECOG Performance status 0-1
* A minimum life expectancy of 12 weeks
* Adequate bone marrow, hepatic and renal function as evidenced by

  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * Hemoglobin > 9.0 g/dL
  * Serum bilirubin < 1.5 x ULN
  * AST/ALT (SGOT/SGPT) < or = 2.5 x ULN for the reference laboratory or < 5 x ULN in the presence of liver metastases
  * Serum creatinine < or = 1.5 x ULN
  * Follicle-Stimulating Hormone (FSH) within normal baseline levels
  * Male patients should have a detectable level of testosterone
* Female patients who are known to be capable of conception should have a negative serum pregnancy test (beta-human chorionic gonadotropin β-hCG]) within 1 week of starting the study.
* All potentially fertile patients will agree to use an effective form of contraception during the study and for 90 days following the last dose of ME-143 (an effective form of contraception is defined as an oral contraceptive or a double barrier method).
* At least 4 weeks must have elapsed prior to Day 1 Cycle 1 since prior chemotherapy (6 weeks for carmustine or mitomycin C), investigational drug or biologic therapy and any toxicity associated with these treatments has recovered to ≤ NCI-CTCAE Grade 1.
* At least 21 days must have elapsed prior to Day 1 Cycle 1, radiotherapy (limited palliative radiation is allowed > 2 weeks), immunotherapy or following major surgery and any surgical incision should be completely healed

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Tumor involvement of the Central Nervous System (CNS) Patients with treated and stable CNS metastases may be eligible to participate after discussion and approval from the Medical Monitor
* Uncontrolled infection or systemic disease.
* Clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease e.g. angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months.
* Patients with QTc of > 470 msec on screening ECG. (If a patient has QTc interval >470 msec on screening ECG, the screening ECG may be repeated twice (at least 24 hours apart). The average QTc from the 3 screening ECGs must be <470 msec in order for the patient to be eligible for the study.
* Any major surgery, radiotherapy, or immunotherapy within the last 21 days (limited palliative radiation is allowed > 2 weeks).
* Chemotherapy regimens with delayed toxicity within the last 4 weeks (or within 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential or delayed toxicity within the last 2 weeks.
* No concurrent systemic chemotherapy or biologic therapy is allowed.
* Known hypersensitivity to any components of ME-143 study drug product.
* Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both).
* History of solid organ transplantation.
* Psychiatric disorder or social or geographic situation that would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | within the first 28 day cycle
  Patients will be administered ME-143 IV infusions weekly and assessed by physical exam, vital signs, hematology and clinical chemistry, urinalysis and pharmacokinetic sampling.

SECONDARY OUTCOMES:
Response rate | baseline and a minimum of every 12 weeks
  radiologic assessments will be performed at baseline and a minimum of every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Mass, MD, Study Chair — MEI Pharma, Inc.
Locations (2):
- United States (2):
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- See also: Sponsor's web site — http://marshalledwardsinc.com
- See also: manuscript — http://link.springer.com/article/10.1007/s10637-013-9949-4